CLINICAL TRIAL: NCT04345666
Title: A Randomized, Blinded Controlled Trial to Determine if Testosterone Can Accelerate Injury Recovery After Arthroscopic Rotator Cuff Repair
Brief Title: Can Testosterone Accelerate Injury Recovery After Arthroscopic Rotator Cuff Repair
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unable to obtain funding to complete the study
Sponsor: Orthopedic Institute, Sioux Falls, SD (Other)
Responsible Party: Principal Investigator, Keith Baumgarten, Orthopedic Surgeon - Physician Scientis, Orthopedic Institute, Sioux Falls, SD
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Orthopedicinstitutesf
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Rotator Cuff Tears
Keywords: arthroscopic rotator cuff repair; testosterone; accelerate recovery from surgery
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — testosterone 17 beta-cypionate

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo controlled model
Who Masked: Participant, Investigator
Masking Description: The patient and the primary investigator will be blinded to the treatment allocation. The study coordinator will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Testosterone group (Experimental): 20 patients will receive a 200 mg testosterone cyprionate intramuscular injection weekly with the first dose started two weeks prior to surgery and the last dose injected at 6 weeks after surgery (9 doses).
  Interventions: Drug: Testosterone cypionate
- Placebo group (Placebo Comparator): 20 patients will receive a sterile saline intramuscular injection weekly with the first dose started two weeks prior to surgery and the last dose injected at 6 weeks after surgery (9 doses).
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Testosterone cypionate — The intervention of this study is to treat patients to either 1) testosterone cypionate or 2) placebo (sterile saline) to determine if there is a difference in recovery times after arthroscopic rotator cuff repair
  Arms: Testosterone group
Drug: Placebos — The intervention of this study is to treat patients to either 1) testosterone cypionate or 2) placebo (sterile saline) to determine if there is a difference in recovery times after arthroscopic rotator cuff repair
  Other Names: Sterile saline
  Arms: Placebo group

SUMMARY:
The objective of this study is to determine if treating patients undergoing arthroscopic rotator cuff repair with testosterone will allow patients to accelerate their recovery time after surgery.

DETAILED DESCRIPTION:
Specific Aim I:

To determine if testosterone treatment would provide superior patient-determined quality-of-life and activity scores in patients undergoing arthroscopic rotator cuff repair compared to a control group at 3 months after surgery.

Specific Aim II:

To determine if testosterone treatment would allow for greater postoperative strength improvements in patients undergoing arthroscopic rotator cuff repair compared to a control group at 3 months after surgery.

Specific Aim III:

To determine if testosterone treatment would allow for greater postoperative range of motion improvements in patients undergoing arthroscopic rotator cuff repair compared to a control group at 3 months after surgery.

Specific Aim IV:

To determine if the potentially higher activity levels allowed by the testosterone treatment would affect the success of rotator cuff healing as determined by magnetic resonance imaging at one year after arthroscopic rotator cuff repair.

The hypothesis of this study was that testosterone treatment of patients undergoing arthroscopic rotator cuff repair would allow patients to achieve 1) better quality-of-life and higher activity levels as determined by patient-determined outcome scores, 2) greater improvements in strength, and 3) greater improvements in range of motion at three months after surgery as compared to the control group. In addition, the authors hypothesize that there would be equivalent healing rates at one year after rotator cuff repair as determined by magnetic resonance imaging between the testosterone group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Males
* arthroscopic rotator cuff repair is an indicated treatment

Exclusion Criteria:

* female patients
* irreparable rotator cuff tears
* tears requiring margin convergence repair
* atrophy of the rotator cuff greater than stage II as determined by the modified Goutallier staging system
* revision rotator cuff repair
* inflammatory arthritis
* adhesive capsulitis
* significant cervical pain or radiculopathy
* history of prostate cancer
* history of benign prostatic hypertrophy
* history of heart failure
* history of obstructive sleep apnea
* history of polycythemia
* history of venous thromboembolism or inherited thrombophilia

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Score | 3 months after surgery
  A validated joint specific patient-determined outcome score (low 0 - 100 high)
American Shoulder and Elbow Score | 6 months after surgery
  A validated joint specific patient-determined outcome score (low 0 - 100 high)
American Shoulder and Elbow Score | 12 months after surgery
  A validated joint specific patient-determined outcome score (low 0 - 100 high)
Simple Shoulder Test | 3 months after surgery
  A validated joint specific patient-determined outcome score (low 0 - 12 high)
Simple Shoulder Test | 6 months after surgery
  A validated joint specific patient-determined outcome score (low 0 - 12 high)
Simple Shoulder Test | 12 months after surgery
  A validated joint specific patient-determined outcome score (low 0 - 12 high)
Single Alpha-Numeric Assessment Evaluation | 3 months after surgery
  A validated general patient-determined outcome score (low 0 - 100 high)
Single Alpha-Numeric Assessment Evaluation | 6 months after surgery
  A validated general patient-determined outcome score (low 0 - 100 high)
Single Alpha-Numeric Assessment Evaluation | 12 months after surgery
  A validated general patient-determined outcome score (low 0 - 100 high)
Shoulder Activity Level | 3 months after surgery
  A validated shoulder-specific activity score (low 0 - 20 high)
Shoulder Activity Level | 6 months after surgery
  A validated shoulder-specific activity score (low 0 - 20 high)
Shoulder Activity Level | 12 months after surgery
  A validated shoulder-specific activity score (low 0 - 20 high)
Shoulder Range of Motion | 3 months after surgery
  Goniometrically-measured (in degrees) Flexion, extension, abduction, external rotation, abducted external rotation, abducted internal rotation, internal rotation behind the back
Shoulder Range of Motion | 6 months after surgery
  Goniometrically-measured (in degrees) Flexion, extension, abduction, external rotation, abducted external rotation, abducted internal rotation, internal rotation behind the back
Shoulder Range of Motion | 12 months after surgery
  Goniometrically-measured (in degrees) Flexion, extension, abduction, external rotation, abducted external rotation, abducted internal rotation, internal rotation behind the back
Shoulder strength | 3 months after surgery
  Dynanometrically measured scaption and external rotation strength (Newtons)
Shoulder strength | 6 months after surgery
  Dynanometrically measured scaption and external rotation strength (Newtons)
Shoulder strength | 12 months after surgery
  Dynanometrically measured scaption and external rotation strength (Newtons)

SECONDARY OUTCOMES:
Magnetic resonance imaging shoulder | 12 months after surgery
  MRI

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Baumgarten, MD, Principal Investigator — Orthopedic Institute
Locations (1):
- Orthopedic Institute, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No
At this point there is no plan to share individual participant data with researcher external to this study